CLINICAL TRIAL: NCT05225714
Title: Assessment of Performance of Silkam® Suture Material for Skin Closure - a Prospective, Single Center, Single Arm, Observational Study in Daily Practice
Brief Title: Dermal Wound Closure Using Silkam®
Acronym: DERMASILK
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1929
Record Dates: First submitted 2022-01-26; First posted 2022-02-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Contusions; Incision; Laceration
MeSH Terms: conditions — Contusions; Surgical Wound; Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of performance of Silkam® suture material for skin closure. A prospective, single center, single arm, observational study in daily practice.

DETAILED DESCRIPTION:
The prospective, monocentric, single-arm, observational Post Market Clinical Follow-Up (PMCF) study is done to continue to evaluate the safety and performance of Silkam® suture material for skin closure under clinical routine. Safety and effectiveness parameters commonly used in skin closure are to be used to evaluate the performance of the suture material.

The aim of this Non Interventional Study is to collect systematically and proactively different clinical parameters regarding safety, effectiveness and performance of Silkam® suture material under the daily routine clinical practice when used for skin closure as intended.

ELIGIBILITY:
Inclusion Criteria:

* Adult and paediatric patients undergoing skin closure using Silkam® as suture material.
* Written informed consent regarding the data collection for the PMCF study.

Exclusion Criteria:

* Pregnancy
* Visible dirty wounds
* Patients taking medication that might affect wound healing
* Patients with hypersensitivity or allergy to the suture material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and paediatric patients undergoing skin closure
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Rate | at suture removal approx. 10 ± 5 days postoperative
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be superficial infections involving the skin only (A1). Other surgical site infections are more serious and can involve tissues under the skin, organs, or implanted material. (A2)

SECONDARY OUTCOMES:
Individual A1 Surgical Site Infection Rate | at suture removal approx. 10 ± 5 days postoperative
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be superficial infections involving the skin only (A1).
Individual A2 Surgical Site Infection Rate | at suture removal approx. 10 ± 5 days postoperative
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be more serious and can involve tissues under the skin, organs, or implanted material. (A2)
Adverse Event Rate | at suture removal approx. 10 ± 5 days postoperative
  frequency of wound dehiscence, hypertrophic scar, keloid scar, inflammation, tissue reaction, seroma, abscess formation, hematoma, granuloma, bleeding, necrosis, skin stripping or irritation.
Cosmetic Outcome | at suture removal approx. 10 ± 5 days postoperative
  Overall patient and observer satisfaction with the scar using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic result and the scar will be evaluated by the patient and the physician. Patient will rate the cosmetic outcome in six categories (Pain, Itching, Color of scar, Stiffness of scar, thickness and irregularity of scar) on a 1 to 10 points scale each. The physician will use the Observer component, rating vascularization, pigmentation, thickness, relief and pliability of the scar on a 1 to 10 points scale each. The categories are added to a total POSAS score of 11 (minimum) to 110 points (maximum).
Pain: Visual Analogue Scale (VAS) | at suture removal approx. 10 ± 5 days postoperative
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".
Satisfaction of the patient: Visual Analogue Scale (VAS) | at suture removal approx. 10 ± 5 days postoperative
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "very poor" and "100" at the opposite end representing "excellent".
Assessment of the handling of the suture material | intraoperative
  Assessment of the handling of the suture material intra-operatively using a questionnaire including different dimensions (knot security, tensile strength, knot run down, tissue drag, pliability) with 5 evaluation levels (excellent, very good, good, satisfied, poor).

OTHER OUTCOMES:
Individual A1 and A2 Surgical Site Infection Rate | at optional follow-up approx. 3 month postoperative
  A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. Surgical site infections can sometimes be superficial infections involving the skin only. Other surgical site infections are more serious and can involve tissues under the skin, organs, or implanted material.
Adverse Event Rate | at optional follow-up approx. 3 month postoperative
  frequency of wound dehiscence, hypertrophic scar, keloid scar, inflammation, tissue reaction, seroma, abscess formation, hematoma, granuloma, bleeding, necrosis, skin stripping or irritation.
Cosmetic Outcome | at optional follow-up approx. 3 month postoperative
  Overall patient and observer satisfaction with the scar using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic result and the scar will be evaluated by the patient and the physician. Patient will rate the cosmetic outcome in six categories (Pain, Itching, Color of scar, Stiffness of scar, thickness and irregularity of scar) on a 1 to 10 points scale each. The physician will use the Observer component, rating vascularization, pigmentation, thickness, relief and pliability of the scar on a 1 to 10 points scale each. The categories are added to a total POSAS score of 11 (minimum) to 110 points (maximum).
Pain: Visual Analogue Scale (VAS) | at optional follow-up approx. 3 month postoperative
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain".
Satisfaction of the patient: Visual Analogue Scale (VAS) | at optional follow-up approx. 3 month postoperative
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "very poor" and "100" at the opposite end representing "excellent".

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Spain